CLINICAL TRIAL: NCT04997382
Title: Chemotherapy Combined with Immune Checkpoint Inhibitors in Patients with ALK-rearranged Non-small Cell Lung Cancer (NSCLC) Who Have Progressed After First-line Alectinib: a Proof-of-concept, Phase 2 Trial
Brief Title: Chemotherapy Combined with ICIs in First-line Alectinib Failed Patients with ALK-rearranged NSCLC
Acronym: CLASSIC5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALICE
Record Dates: First submitted 2021-07-31; First posted 2021-08-09 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Alectinib; ALK Rearranged
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immune Checkpoint Inhibitors; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Based on the treatment preferences of each patient, they received either chemotherapy alone or in combination with immune checkpoint inhibitors, as well as chemotherapy in combination with immune checkpoint inhibitors (ICI), either with or without bevacizumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Patients with 3'ALK retained 5'ALK. (Experimental): Patients with 3'ALK retained 5'ALK who progressed from first line Alectinib were randomized to Arm A: Chemo+ICIs/Chemo+ICIs+BEV and Arm B: Chemo/Chemo+BEV.
  Interventions: Drug: Chemotherapy alone or Chemotherapy plus Immune Checkpoint Inhibitors with or without Bevacizumab; Drug: Chemotherapy alone or Chemotherapy with or without Bevacizumab
- Part B: Patients with 3'ALK. (Experimental): Patients with 3'ALK who progressed from first line Alectinib were randomized to Arm C: Chemo+ICIs/Chemo+ICIs+BEV and Arm D: Chemo/Chemo+BEV.
  Interventions: Drug: Chemotherapy alone or Chemotherapy plus Immune Checkpoint Inhibitors with or without Bevacizumab; Drug: Chemotherapy alone or Chemotherapy with or without Bevacizumab

INTERVENTIONS:
Drug: Chemotherapy alone or Chemotherapy plus Immune Checkpoint Inhibitors with or without Bevacizumab — Immune Checkpoint Inhibitors, for pembrolizumab, 200mg ivgtt once,every 21 days; for Atezolizumab, 1200mg vgtt once,every 21 days.
  Other Names: Bevacizumab
Drug: Chemotherapy alone or Chemotherapy with or without Bevacizumab — Bevacizumab, 15mg/kg，every 21 day
  Other Names: Bevacizumab

SUMMARY:
This study aimed to investigate the combination of chemotherapy and immunotherapy for patients with metastatic ALK fusion-positive non-small cell lung cancer (NSCLC) who had failed from first line Alectinib. Additionally, available biological samples such as blood and tumor tissues were collected to explore potential biomarkers, including but not limited to RNA-seq, whole-exome sequencing (WES), whole-genome sequencing (WGS), immunohistochemistry, and multiplex immunofluorescence.

DETAILED DESCRIPTION:
1. The investigators collected data from patients with metastatic ALK fusion-positive non-small cell lung cancer (NSCLC) who received first-line Alectinib treatment between April 2017 and July 2021. Our analysis aimed to assess their clinical outcomes and explore the impact of 5' ALK on the treatment response to Alectinib.
2. For patients who experienced disease progression after August 2021, they were treated with a combination of chemotherapy and PD-1 monoclonal antibodies with/without Bevacizumab or chemotherapy alone with/without Bevacizumab was observed and recorded data on progression-free survival (PFS), objective response rate (ORR), duration of response (DOR), and overall survival (OS) for these patients.
3. The investigators collected pre-treatment biological samples for biomarker analysis, including FFPE samples for whole-genome sequencing (WGS), whole-exome sequencing (WES), RNA-seq, and multiplex fluorescence analysis. FFPE samples were also collected for PD-L1 testing. Additionally, pre-treatment blood samples were collected for cytokine analysis, as well as tumor mutational burden (TMB) and T-cell receptor (TCR) testing. The investigators aimed to evaluate the differences in these results between 3' ALK and 5' ALK.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18，Advanced Non-small Cell Lung Cancer Confirmed by Histopathology
2. ALK -arreaged confirmed by NGS;
3. Received first line treatment Alectinib;
4. Progressed from first-line alectinib;
5. ECOG 0-1;
6. Predicted survival ≥ 12 weeks;
7. Adequate bone marrow hematopoiesis and organ function;
8. Presence of measurable lesions according to RECIST 1.1;
9. Subjects with stable brain metastases may be included in the study.
10. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.

Exclusion Criteria:

1. Patient who do not have the samples for NGS to confirmed ALK status.
2. Subjects who have received any of the following treatments must be excluded:

   * Treatment with molecules such as EGFR, VEGFR antibodies within 4 weeks prior to the first dose of study drug.
   * Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
3. Presence of spinal cord compression or meningeal metastasis.
4. History of other malignant tumors within 2 years.
5. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
6. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
7. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
8. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
9. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb sunvozertinib or anlotinib due to previous bowel resection.
10. Live vaccine was given 2 weeks before the first medication.
11. Women who are breastfeeding or pregnant.
12. Hypersensitivity to the test drug and the ingredients.
13. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
PFS | From first dose until 28 days after the last dose, up to 24 months
  Progression free survival time

SECONDARY OUTCOMES:
OS | Time from first subject dose to study completion, or up to 48 months
  Overall survival time
ORR | From first dose until 28 days after the last dose, up to 24 months
  Objective Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No